CLINICAL TRIAL: NCT05360381
Title: A Phase I Clinical Study Evaluating the Safety, Tolerability, Pharmacokinetic Characteristics and Initial Efficacy of HLX35 (Recombinant Human Anti-EGFR and Anti-4-1BB Bispecific Antibody) in Patients With Advanced or Metastatic Solid Tumors
Brief Title: HLX35(EGFR×4-1BB Bispecific) in Patients With Advanced or Metastatic Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HLX35-FIH101
Record Dates: First submitted 2022-04-26; First posted 2022-05-04 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Locally Advanced or Metastatic Solid Tumors; Squamous-cell Non-small Cell Lung Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase 1a dose-escalation stage (Experimental): Phase 1a uses the "3+3" design, to investigate the safety and determine the MTD of HLX35. Seven dose levels of 0.015 mg/kg, 0.05 mg/kg, 0.1 mg/kg, 0.3 mg/kg, 1 mg/kg, 3 mg/kg, and 10 mg/kg are planned for dose finding. Enrollment will continue until a maximum of 42 patients are enrolled
  Interventions: Drug: HLX35
- Phase 1b dose-expansion stage (Experimental): Patients with sqNSCLC (EGFR H score≥200) will be enrolled in two expansion cohorts, at doses equal to or lower than the MTD, to better characterize the safety, tolerability, PK variability, and preliminary efficacy of single-agent HLX35. Phase 1b dose expansion will include 15-20 per-protocol treated patients, as defined above, in each of the two expansion cohorts.
  Interventions: Drug: HLX35

INTERVENTIONS:
Drug: HLX35 — A Recombinant Human Anti-EGFR and Anti-4-1BB Bispecific Antibody, HLX35 will be administered as a single intravenous (IV) infusion on Day 1 in each 14-day cycle

SUMMARY:
This Phase1, multicenter, first-in-human, open-label, dose-escalation, and dose expansion study will evaluate the safety, tolerability, pharmacokinetics, and preliminary anti-tumor efficacy of HLX35 administered as a single-agent by IV infusion every 2 weeks to patients with locally advanced or metastatic solid malignancies, who have failed or are intolerant to standard therapy, or for whom no standard therapy is available. This study has two parts: phase 1a dose escalation and phase 1b dose expansion.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in this clinical study; completely understand and know this study as well as sign the informed consent form (ICF);
* Age ≥ 18 years;
* Phase 1a dose escalation: patients must have histologically or cytologically confirmed malignant solid tumors which are advanced or metastatic, have failed prior standard treatment, and be intolerant or ineligible for standard therapy;
* Phase 1b dose expansion: patients must have a histological or cytological diagnosis of Squamous Non-Small Cell Lung Cancer (EGFR H score ≥200 confirmed by central lab) which is advanced or metastatic, have failed prior standard treatment, and be intolerant or ineligible for standard therapy;
* Measurable disease according to RECIST Version 1.1;
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1;
* Expected survival 12 weeks;
* Adequate organ function;

Exclusion Criteria:

* Systemic anti-cancer treatment or investigational agents in the 28 days prior to the first study dosing;
* Patients who still have persistent ≥ grade 2 toxicities from prior therapies;
* Active CNS metastasis;
* History of any secondary malignancy in the past 5 years;
* Active autoimmune disease;
* Human immunodeficiency virus (HIV) infection;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2022-06-03 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Related Adverse Events | 2 years
The proportion of patients experiencing dose limiting toxicity (DLT) events | from first dose to the end of Cycle 2 (each cycle is 14 days)
The maximum tolerated dose (MTD) | from first dose to the end of Cycle 2 (each cycle is 14 days)
Recommended phase 2 dose (RP2D) | from first dose to the end of Cycle 2 (each cycle is 14 days)

SECONDARY OUTCOMES:
Peak plasma concentration (Cmax) of HLX35 | 2 years
Time to peak (Tmax) of HLX35 | 2 years
Area under the concentration-time curve (AUC) of HLX35 | 2 years
Elimination half-life (t1/2) of HLX35 | 2 years
Clearance (CL) of HLX35 | 2 years
Volume of distribution (Vz) of HLX35 | 2 years
Accumulation Index (Rac) of HLX35 | 2 years
4-1BB receptor occupancy on circulating T cells | 2 years
The level of 4-1BB in serum | 2 years
Incidence of treatment-emergent anti-drug antibodies (ADA) | 2 years
Objective response rate (ORR) | 2 years
Disease control rate (DCR) | 2 years
Duration of response (DOR) | 2 years

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Fudan University Shanghai Cancer Center, Shanghai
  - THE Affiliated Hospital of Xuzhou Medical University, Xuzhou

IPD SHARING:
Plan to Share IPD: Undecided